CLINICAL TRIAL: NCT02160951
Title: A Multi-center, Open-label, Dose Escalation, Phase 1 Study of Oral LGH447 in Japanese Patients With Relapsed and/or Refractory Hematologic Malignancies
Brief Title: Dose Escalation Study of LGH447 in Japanese Patients With Relapsed and/or Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLGH447X1101
Record Dates: First submitted 2014-05-30; First posted 2014-06-11 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2017-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma,; Phase I,; PIM,; Japanese patients,; LGH447
MeSH Terms: conditions — Multiple Myeloma | interventions — LGH-447

ARMS (1):
- LGH447 (Experimental): LGH447, QD
  Interventions: Drug: LGH447

INTERVENTIONS:
Drug: LGH447 — LGH447, QD

SUMMARY:
This is a multi-center, open-label, dose escalation, Phase 1 study of oral LGH447 in Japanese patients with relapsed and/or refractory multiple myeloma for which no standard effective treatment options exist.

The study consists of a dose escalation part to estimate the maximum tolerated dose and/or the recommended dose for expansion and a dose expansion part to further assess safety and preliminary anti-cancer activity of LGH447 at the maximum tolerated dose and/or the recommended dose for expansion.

ELIGIBILITY:
Inclusion Criteria:

-Confirmed diagnosis of relapsed and/or refractory MM for which no standard effective treatment options exist.

Exclusion Criteria:

-Uncontrolled cardiovascular condition, including ongoing cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence rate of dose limiting toxicities | 28 days
  Estimate the maximum tolerated dose and/or recommended dose for expansion of LGH447 in Japanese patients

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability of LGH447 | 28 days and till the end of the study, an average of 84 days
  Adverse events, serious adverse events, changes in laboratory values, and electrocardiograms
Pharmacokinetics profile of LGH447 and its metabolites if appropriate | Baseline, 0.5, 1, 2, 3, 4, 5, 6, 8, 24 hours on Cycle1Day1, 14 and 28 and baseline on Cycle2Day14 and Cycle3Day1
  PK parameters such as AUC, Cmax, Tmax, T1/2. Cycle = 28 days
Overall Response Rate | Every 28 days till the end of the study, an average of 84 days
  Describe any preliminary anti-cancer activity associated with LGH447 based on International Myeloma Working group Criteria with modification.
Disease control rate | Every 28 days till the end of the study, an average of 84 days
  Describe any preliminary anti-cancer activity associated with LGH447 based on International Myeloma Working group Criteria with modification.
Clinical benefit rate | Every 28 days till the end of the study, an average of 84 days
  Describe any preliminary anti-cancer activity associated with LGH447 based on International Myeloma Working group Criteria with modification.
Duration of Response | Every 28 days till the end of the study, an average of 84 days, from the first documented onset of confirmed PR or better response to the date of documented disease progression/relapse or death due to multiple myeloma
  Describe any preliminary anti-cancer activity associated with LGH447 based on International Myeloma Working group Criteria with modification.
Progression Free Survival | Every 28 days till the end of the study, an average of 84 days, from start of treatment to the date of event defined as the first documented disease progression/relapse, or death due to any cause
  Describe any preliminary anti-cancer activity associated with LGH447 based on International Myeloma Working group Criteria with modification.
Time to response | Every 28 days till the end of the study, an average of 84 days, from start of treatment until first documented best overall response
  Describe any preliminary anti-cancer activity associated with LGH447 based on International Myeloma Working group Criteria with modification.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Japan (4):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Okayama, Okayama-ken

REFERENCES:
- [Derived] Iida S, Sunami K, Minami H, Hatake K, Sekiguchi R, Natsume K, Ishikawa N, Rinne M, Taniwaki M. A phase I, dose-escalation study of oral PIM447 in Japanese patients with relapsed and/or refractory multiple myeloma. Int J Hematol. 2021 Jun;113(6):797-806. doi: 10.1007/s12185-021-03096-9. Epub 2021 Feb 27. PMID 33638035
- See also: Results for CLGH447X1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=15748